CLINICAL TRIAL: NCT02817360
Title: NT-proBNP Selected PreventiOn of Cardiac eveNts in a populaTion of dIabetic Patients Without A History of Cardiac Disease: a Prospective Randomized Trial
Brief Title: NT-proBNP Selected Prevention of Cardiac Events in Diabetic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Martin Huelsmann (Other)
Responsible Party: Sponsor-Investigator, Martin Huelsmann, Univ.Doz. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PONTIAC II
Record Dates: First submitted 2016-02-15; First posted 2016-06-29 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Heart Diseases; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus, Type 2 | interventions — Enalapril; Ramipril; Lisinopril; Cilazapril; Perindopril; Captopril; spirapril; Quinapril; trandolapril; zofenopril; Fosinopril; candesartan; Valsartan; Irbesartan; Losartan; eprosartan; Bisoprolol; Carvedilol; Nebivolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive therapy (Experimental): RAS-antagonist and beta-blocker up-to maximal dosages as permitted and tolerated and following national guidelines.
  Interventions: Drug: RAS-antagonist and beta-blocker up-to maximal dosages
- Conventional therapy (Other): No RAS-antagonist and beta-blocker or at stable dose as per study entrance. Changes in RAS-antagonist or beta-blocker therapy are not allowed in the control group during the study phase.
  Interventions: Other: RAS-antagonist and beta-blocker none or at stable dose

INTERVENTIONS:
Drug: RAS-antagonist and beta-blocker up-to maximal dosages — All patients have to be stable on their glucose lowering, lipid lowering and blood pressure lowering therapy at least for 3 months. RAS-antagonist and beta-blocker therapy at entrance is allowed. Patients receive a prescription and/or up-titration to maximum recommended or tolerated dose of RAS-antagonist and beta-blockers within three months of study entry. The Number of titration visits is up to the treating physician, but one visit should be performed at least at the end of titration.
  Other Names: Enalapril 40mg/d; Ramipril 10mg/d; Lisinopril 40mg/d; Cilazapril 5mg/d; Perindopril 8mg/d; Captopril 150mg/d; Spirapril 24mg/d; Quinapril 40mg/d; Trandolapril 4mg/d; Zofenopril 60mg/d; Fosinopril 40mg/d; Candesartan 32mg/d; Valsartan 320mg/d; Irbesartan 300mg/d; Losartan 150mg/d; Eprosartan 800mg/d; Bisoprolol 10mg/d; Metoprololsuccinat 200mg/d; Carvedilol 50mg/d (100mg/d if weight is > 85kg); Nebivolol 10mg/d
  Arms: Intensive therapy
Other: RAS-antagonist and beta-blocker none or at stable dose — All patients have to be stable on their glucose lowering, lipid lowering and blood pressure lowering therapy at least for 3 months. RAS-antagonist and beta-blocker therapy at entrance is allowed. Changes in RAS-antagonist or beta-blocker therapy are not allowed in the control group during the study phase. If there is a vital indication for changes, this has to be argued and documented.
  Arms: Conventional therapy

SUMMARY:
Purpose and rationale The purpose of this study is to evaluate the effect of high dose Renin-Angiotensin System (RAS)-antagonists and beta-blocker treatment for the primary prevention of cardiac events in a population of patients with Type 2 diabetes mellitus (T2DM) with no evidence of a preexisting cardiac disease. An additional aim is to demonstrate an interaction between concentrations of amino-terminal pro-B type natriuretic peptide (NT-proBNP as a surrogate of imminent cardiac risk) and treatment effects and the economic impact of the intervention overall and in the biomarker stratified subgroups.

Primary objective Superiority of high dose treatment with RAS-antagonists and beta-blockers compared to conventional therapy regarding the reduction of unplanned hospitalization or death due to a cardiac event in T2DM patients with a NT-proBNP > 125pg/ml.

There is an additional eye-substudy for Viennese sites only. The purpose of this sub-study is to evaluate the effect of high dose RAS-antagonists and beta blocker treatment on early subclinical signs of diabetic micro-angiopathy and neuropathy. An additional aim will be the evaluation of the possible impact of the cardiovascular risk factor NT-proBNP on the onset and progression of diabetic retinopathy.

DETAILED DESCRIPTION:
Purpose and rationale The purpose of this study is to evaluate the effect of high dose Renin-Angiotensin System (RAS)-antagonists and beta-blocker treatment for the primary prevention of cardiac events in a population of patients with Type 2 diabetes mellitus (T2DM) with no evidence of a preexisting cardiac disease. An additional aim is to demonstrate an interaction between concentrations of amino-terminal pro-B type natriuretic peptide (NT-proBNP as a surrogate of imminent cardiac risk) and treatment effects and the economic impact of the intervention overall and in the biomarker stratified subgroups.

Primary objective Superiority of high dose treatment with RAS-antagonists and beta-blockers compared to conventional therapy regarding the reduction of unplanned hospitalization or death due to a cardiac event in T2DM patients with a NT-proBNP > 125pg/ml.

Co-primary objective Superiority of high dose treatment with RAS-antagonists and beta-blockers compared to conventional therapy regarding the reduction of unplanned hospitalization or death due to a cardiac event in T2DM patients in the whole population Secondary objective Dependency of treatment efficacy (reduction of unplanned hospitalization or death due to a cardiac event in T2DM patients) on the NT-proBNP concentration (interaction effect between NT-proBNP concentrations and treatment).

Population The study population will consist of patients with T2DM without any history or signs of cardiac disease. Patients from approximately 20 centers worldwide will be included into the study and randomized 1:1 to intensive or conventional therapy. It is estimated that about 3000 patients have to be screened In order to include 2400 patients. The screen failure rate is anticipated to be approximately 20%.

Investigational and reference therapy All eligible patients will be randomized to receive either a high dose of RAS-antagonists and beta-blockers (as defined in the section investigational drugs) on top of standard diabetes therapy or solely standard diabetes therapy. The use of RAS-antagonist and beta-blocker therapy at randomization is allowed in the control group (with the exception of maximal dosage), but prescription or titration during the study period is not encouraged. However, if the investigators feel that further prescription or up-titration is required a thorough justification is mandatory. Every attempt should be made to use other blood pressure lowering drugs than RAS-antagonists or beta-blockers in the control group.

Study design This study is a randomized open-label, parallel group, active-controlled, two-arm, long-term morbidity and mortality trial to evaluate the efficacy and safety of high dose RAS-antagonist and beta-blocker therapy (as defined in the section investigational drugs) compared to standard diabetes therapy in patients with diabetes without any history or sign of a cardiac disease.

The goal is to include 2400 patients. The observation period is planned to last for two years. However, the trial is event driven and will continue until predefined event rate is reached. The total trial duration is expected to last for four years (two years of recruitment and a two year observation period after last patient in). Every patient will remain in the study for two years after randomization.

Visit 1 Screening At the first visit eligibility to enter the study will be assessed by the investigator. All inclusion/exclusion criteria will be evaluated. Informed consent will be obtained. Demographic data and drug prescription will be assessed. Blood will be obtained. Blood chemistry will be assessed locally. NT-proBNP will be determined by a point of care system locally. The investigator will be blinded to the result, which will be sent to the central computer. Blood will be obtained for the core lab, centrifuged and stored at -80° Celsius at the local unit. Vital signs will be obtained. Randomization will be performed electronically, this way randomization can be performed immediately.

Visit 2 (3 months) At visit 2 vital signs will be obtained. Blood will be drawn. Blood chemistry parameters will be assessed locally for safety reason. Drug prescription will be documented.

Visit 3 (12 months) At visit 3 vital signs will be obtained. Blood will be drawn. Blood chemistry parameters will be assessed locally for safety reason. Drug prescription will be documented.

Visit 4 EOS (end of study) (24 months) At visit 4 vital signs will be obtained. Blood will be drawn. Blood chemistry parameters will be assessed locally for safety reason. Additional blood samples will be sent to the core laboratory. Drug prescription will be documented.

Visit 1-4 is mandatory for all patients. Long-term follow-up Patients with be further followed by population register or telephone contact respectively until completion of the study to determine long-term mortality and hospitalizations.

Unscheduled visits for the treatment group The treatment group will have additional visits for up-titration of RAS-antagonists and beta- blocker between visit 1 and visit 2. The frequency is up to the treating physician and dependent on the titration steps. A visit is not mandatory for each titration step. Patients will receive a logbook by the investigator, with weekly up- titration steps of the drugs. Additionally, patients will receive a diary for daily documentation of blood pressure, heart rate and symptoms if measurement is technically feasible for the patient. Based on own measurements, these data and laboratory results the investigator will decide if further up-titration of medication is possible. Systolic blood pressure should not decrease permanently below 100 mmHg and heart not below 60bpm permanently. Recommended drugs and recommended dosages are outlined in the section "Treatment". At each visit, blood chemistry for eGFR, creatinine, blood urea nitrogen (BUN), sodium and potassium will be obtained for safety reason.

Details of the eye-substudy:

The PONTIAC Eye Study is a masked longitudinal follow up of previously 1:1 randomized study patients participating in the PONTIAC 2 study. It is planed to include 130 consecutive patients for biannually visits over a study period of 2 years. Study patients (n=130) will be assigned to the Department of Ophthalmology and Optometry of the Medical University Vienna once they are included in the PONTIAC 2 Study in one of the participating Centers in Vienna. The investigators will be masked to the patient's randomization.

The primary objective of the sub-study is: Superiority of the treatment arm with RAS-antagonists and beta-blockers compared to conventional therapy regarding thickness-change in the retinal nerve fiber layer or outer nuclear layer measured in spectral domain optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

1. Type-2 diabetes for at least six months,
2. ≥ 18 years of age, men or female,
3. Written informed consent to participate in the study and ability to comply with all requirements.

Exclusion Criteria:

1. History of hypersensitivity to any of the investigated drugs as well as known or suspected contraindications to the study drugs or previous history of intolerance to high dose of RAS-Antagonist or Beta-blocker in the absence of any other blood pressure lowering drugs.
2. Patients already on maximum dose of RAS-antagonist or beta-blocker.
3. Creatinine > 2.5mg/dl.
4. Symptomatic hypotension and/or systolic blood pressure (SBP) < 100 mmHg at Visit 1.
5. Symptomatic bradycardia and/or heart rate (HR) < 60 bpm at Visit 1
6. Signs of cardiac disease in the ECG such as atrial fibrillation; ST-T abnormalities or any bundle branch block / higher degree atrioventricular (AV) block.
7. Abnormal echocardiography, defined as low ejection fraction < 50%; wall motion abnormalities suggesting coronary artery disease (CAD), significant valve dysfunction > grade I or other significant alteration.
8. Coronary artery disease, defined by a history of myocardial infarction, known coronary stenosis > 70% detected either by angiography or by CT-scan, significant defects in myocardial scintigraphy or positive stress-test echocardiography.
9. A disease other than T2DM lowering the patient's life expectancy to less than two years.
10. Chronic infections or malignancies.
11. Systemic treatment with corticosteroids.
12. Renal replacement therapy.
13. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy OR are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation), hormonal contraception (implantable, patch, and oral), and double-barrier methods (if accepted by local regulatory authority and ethics committee). Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive Human Chorionic Gonadotropin (hCG) laboratory test (> 5 U/ml).
15. History of noncompliance to medical regimes and patients who are considered potentially unreliable.
16. Current double blind treatment in diabetic trials.
17. Participation in an investigational drug study at the time of enrollment or within the past 90 days.

Eligibility criteria for eye-substudy:

Inclusion criteria:

1. Participation in the PONTIAC 2 Study
2. Written informed consent to participate in the eye-study

Exclusion criteria:

1. Media opacities like cataract or vitreous hemorrhage
2. Active intraocular inflammation (grade trace or above) in either eye like infectious conjunctivitis, keratitis, scleritis, endophthalmitis as well as idiopathic or autoimmune-associated uveitis in either eye
3. Structural damage to the center of macula in the study eye
4. Atrophy of retinal pigment epithelium, subretinal fibrosis, laser scar within foveal avascular zone (FAZ) or organized hard exudate plaques
5. Ocular disorders in the study eye including retinal vascular occlusion, retinal detachment, macular hole, choroidal neovascularization, macula dystrophies
6. Intraocular surgery (including cataract surgery, Yttrium-Aluminium-Granat (YAG) laser capsulotomy) in the study eye within 3 months preceding Day 0
7. Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication)
8. History of glaucoma filtration surgery, corneal transplantation in the study eye
9. Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded
10. History of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with an unplanned cardiac hospitalization or death due to a cardiac event | 2 years
  The combined endpoint of the number of patients with an unplanned cardiac hospitalization or death due to a cardiac event will be recorded throughout the study duration of 2 years.

OTHER OUTCOMES:
Number of patients hospitalised due to any cardiac reasons | 2 years
  The number of subjects who were hospitalised due to any cardiac reasons will recorded.
Number of patients hospitalised due to heart failure | 2 years
  The number of subjects who were hospitalised due to a heart failure will recorded.
Number of patients hospitalised due to all causes | 2 years
  The number of subjects who were hospitalised due to any cause
Change of kidney function | 2 years
  Change of kidney function measured by eGFR (estimated glomerular filtration rate)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Huelsmann, Doz.Dr., Principal Investigator — Univ.Clinic II, Medical University Vienna
Locations (21):
- Austria (11):
  - Internistische Ordination, Mödling, Lower Austria
  - Klinischen Abteilung für Endokrinologie und Diabetologie MU Graz, Graz, Styria
  - Konventhospital der Barmherzigen Brüder Abteilung für Innere Medizin, Linz, Upper Austria
  - Krankenanstalt Rudolfstiftung, 1. Medizinische Abteilung, Vienna
  - Zentrum für Klinische Studien, Vienna
  - Medical University of Vienna Univ.Clinic for Internal Medicine II Department of Cardiology, Vienna
  - Univ. Klinik für Innere Medizin III Med. Uni Wien, Vienna
  - Universitätsklinik für Augenheilkunde und Optometrie Medizinische Universität Wien, Vienna
  - Diabetes & Stoffwechselambulanz Gesundheitszentrum Wien Süd, Vienna
  - 3. Med. Abtlg., KH Hietzing mit Neurologischem Zentrum Rosenhügel, Vienna
  - iMED19, Vienna
- Maastricht University Medical Center; Dep. Cardiology, Maastricht, Netherlands
- Christchurch Heart Institute, Christchurch, New Zealand
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Unitat de Diabetis, Servei d'Endocrinologia i Nutrició, Universitat Autònoma de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, l'Institut del Cor, Barcelona
- United Kingdom (6):
  - Ninewells Hospital, Diabetes Support Unit, Dundee
  - Queen Elisabeth University Hospital, Glasgow Clinical Research Facility, Glasgow
  - North Manchester General Hospital, Diabetes centre, Manchester
  - Nethergreen Surgery, Sheffield
  - Ecclesfield Group Practice, Sheffield
  - Woodseats Medical Centre, Sheffield

IPD SHARING:
Plan to Share IPD: No